CLINICAL TRIAL: NCT00563056
Title: Open, Randomised, Parallel Group Multicentre Study to Compare the Efficacy & Safety of Flutiform® pMDI vs Fluticasone pMDI Plus Formoterol DPI in Adolescent & Adult Subjects With Mild to Moderate-severe Persistent, Reversible Asthma
Brief Title: An Open, Randomised, Parallel Group Multicentre Study to Compare the Efficacy and Safety of Flutiform® pMDI vs Fluticasone pMDI Plus Formoterol DPI in Adolescent and Adult Subjects With Mild to Moderate-severe Persistent, Reversible Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLT3505; 2007-001634-13
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Asthma Bronchiale
Keywords: Formoterol; Fluticasone; Asthma
MeSH Terms: conditions — Asthma | interventions — fluticasone-formoterol; Fluticasone; Formoterol Fumarate

ARMS (2):
- Flutiform (Experimental): 2 puffs 50/5 or 125/5 mcg
  Interventions: Drug: Flutiform
- Flixotide plus Foradil (Active Comparator): Flixotide 2 puffs 50 or 125 mcg; Foradil 1 puff 12 mcg
  Interventions: Drug: Flixotide plus Foradil

INTERVENTIONS:
Drug: Flutiform
  Arms: Flutiform
Drug: Flixotide plus Foradil
  Arms: Flixotide plus Foradil

SUMMARY:
Flutiform® compared with the individual components Flixotide® (Fluticasone) and Foradil® (Formoterol) in adolescent and adult patients.

DETAILED DESCRIPTION:
This is a study involving a 12 week treatment phase. During the treatment phase subjects receive Flutiform® or Flixotiole® and Foradil® as individual componements. Efficacy will be assessed by lung function tests and asthma symptoms, sleep disturbance. Safety will be assessed by adverse events, vital signs, lab tests and ECGs.

ELIGIBILITY:
Inclusion criteria:

1. Male or female subjects at least 12 years or older (females less than one year post-menopausal must have a negative serum or urine pregnancy test recorded at the screening visit prior to the first dose of study medication, be non-lactating, and willing to use adequate and highly effective methods of contraception throughout the study if they are sexually active. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilization, implants, injectables, combined oral contraceptives, some IUDs (Intrauterine Device, hormonal), sexual abstinence or vasectomised partner).
2. Known history of mild to moderate-severe persistent, reversible asthma for ≥ 6 months prior to the screening visit.
3. Demonstrate a FEV1 of ≥40% to ≤85% for predicted normal values (Quanjer et al, 19931) during the screening phase following appropriate withholding of asthma medications (if applicable).

   * No β2-agonist use on day of screening.
   * No use of inhaled combination asthma therapy on day of screening.
   * Inhaled corticosteroids are allowed on day of screening.
4. Documented reversibility of ≥15% in FEV1 in the screening phase.
5. Demonstrate satisfactory technique in the use of the study medications.
6. Willing and able to enter information in the diary and attend all study visits.
7. Willing and able to substitute study medication for their pre study prescribed asthma medication for the duration of the study.
8. Written informed consent obtained

Exclusion criteria:

1. Near fatal or life-threatening (including intubation) asthma within the past year.
2. Hospitalization or an emergency visit for asthma within the past year.
3. History of systemic (oral or parenteral) corticosteroid medication within 1 month before the Screening Visit.
4. History of omalizumab use within the past 6 months.
5. History of leukotriene receptor antagonist use, e.g. montelukast, or theophylline within the past week.
6. Current evidence or history of any clinically significant disease or abnormality including uncontrolled coronary artery disease, congestive heart failure, myocardial infarction, or cardiac dysrhythmia. 'Clinically significant' is defined as any disease that, in the opinion of the Investigator, would put the patient at risk through study participation, or which would affect the outcome of the study.
7. In the investigators opinion a clinically significant upper or lower respiratory infection within 4 weeks prior to the Screening Visit.
8. Significant, non-reversible, active pulmonary disease (e.g., chronic obstructive pulmonary disease (COPD), cystic fibrosis, bronchiectasis, tuberculosis).
9. Known Human Immunodeficiency Virus (HIV)-positive status.
10. A smoking history equivalent to "10 pack years" (i.e., at least 1 pack of 20 cigarettes /day for 10 years or 10 packs/day for 1 year, etc.).
11. Current smoking history within 12 months prior to the Screening Visit.
12. Current evidence or history of alcohol and/or substance abuse within 12 months prior to the Screening Visit.
13. Subjects who have taken B-blocking agents, tricyclic antidepressants, monoamine oxidase inhibitors, astemizole (Hismanal), quinidine type antiarrhythmics, or potent CYP 3A4 inhibitors such as ketoconazole within the past week.
14. Current use of medications that will have an effect on bronchospasm and/or pulmonary function.
15. Current evidence or history of hypersensitivity or idiosyncratic reaction to test medications or components.
16. Receipt of an investigational drug within 30 days of the Screening Visit (12 weeks if an oral or injectable steroid).
17. Current participation in a clinical study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Comparison of mean Forced Expriatory Volume in the 1st second (FEV1) values. | 12 weeks

SECONDARY OUTCOMES:
Discontinuation, PEFR, rescue medication use, asthma symptom scores, sleep disturbance, AQLQ, exacerbations, patient acceptance | 12 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- Research Site, Kassel, Germany
- Research Site, Érd, Hungary
- Research site, Nieuwegein, Netherlands
- Research Site, Krakow, Poland
- Research Site, Cluj-Napoca, Romania
- Research Site, Chesterfield, United Kingdom

REFERENCES:
- [Derived] Bodzenta-Lukaszyk A, van Noord J, Schroder-Babo W, McAulay K, McIver T. Efficacy and safety profile of fluticasone/formoterol combination therapy compared to its individual components administered concurrently in asthma: a randomised controlled trial. Curr Med Res Opin. 2013 May;29(5):579-88. doi: 10.1185/03007995.2013.772506. Epub 2013 Feb 20. PMID 23368897
- See also: Results available on register — https://www.clinicaltrialsregister.eu/ctr-search/search?query=FLT3505